CLINICAL TRIAL: NCT03562715
Title: Role of Mesenchymal Stem Cells Exosomes Derived microRNAs; miR-136, miR-494 and miR-495 in Pre-eclampsia Diagnosis and Evaluation
Brief Title: microRNAs Role in Pre-eclampsia Diagnosis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadine wagdi maurice, Teaching assistant at biochemistry department Faculty of pharmacy, Cairo University
Other Study IDs: BC (1870)
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Preeclampsia
Keywords: microRNAs; exosomes; preeclampsia; mesenchymal stem cells
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Blood samples were collected from 100 control with normal pregnancies. Thirty fresh umbilical cord samples of women with healthy pregnancies (n=15) were retrieved during caesarean deliveries and umibilical cord mesenchymal stem cells (UCMSCs) were isolated from Wharton jelly.
- Preeclampsia group: Blood samples were collected from 100 patients with PE. Thirty fresh umbilical cord samples of PE patients (n=15) were retrieved during caesarean deliveries and UCMSCs were isolated from Wharton jelly.

SUMMARY:
Pre-eclampsia is one of the most threatening pregnancy complications. So far neither a secure, competent therapy for PE nor effective biomarkers for a premature discovery has been achieved.The aim of our study was to identify miRNAs 136, 494 and 495 genes expression in exosomes of peripheral blood compared to umbilical cord mesenchymal stem cells conditioned media released exososomes in patients with PE, as valuable markers for PE early prediction.

ELIGIBILITY:
Inclusion Criteria:

To have an uncomplicated pregnancy:

1. gestational age at venipuncture between 20 - 42 weeks
2. no medical, obstetrical, or surgical complications
3. absence of labor at the time of venipuncture
4. delivery of a normal term (≥ 37 weeks) neonate whose birth weight was between the 10th and 90th percentile for gestational age

Exclusion Criteria:

Patients with chronic hypertension, renal disease, and fetuses affected with congenital anomalies were excluded

Ages: 23 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: PE group included 100 females with a mean age of 28.77 ± 5.72 years, while control group comprised of 100 females with a mean age of 28.06 ± 5.65 years. All enrolled patients were clinically diagnosed by physical examination and laboratory investigations.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
The expression of miRNAs 136, 494 and 495 in exosomes of peripheral blood and UCMSCs conditioned media | 2-3 months